CLINICAL TRIAL: NCT00197171
Title: Evaluate the Persistence of Immune Response of GSK Biologicals' TWINRIX™ ADULT, Administered According to 0,6 Month Schedule and 0,12 Month Schedule, in Volunteers Aged 12-15 Years Inclusive at the Time of First Vaccine Dose
Brief Title: Long Term F/U Studies at Y5&6 to Demonstrate the Equivalence of 2 Vaccination Schedules of Combined Hepatitis A & B Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100386 (EXT Y5); 100387
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B; Hepatitis A
MeSH Terms: conditions — Hepatitis B; Hepatitis A

INTERVENTIONS:
Biological: Combined Hepatitis A and B vaccine

SUMMARY:
To evaluate the persistence of immune response 5 years and 6 years after the first vaccine dose.

DETAILED DESCRIPTION:
Open, randomised, long-term antibody persistence studies, conducted in 2 centers. Immune persistence was compared between subjects who received two doses of GSK Biologicals combined hepatitis A and hepatitis B vaccine at either 0, 6 month schedule or 0, 12 month schedule. These long-term follow-up studies involved taking blood samples at approximately 5 and 6 years after the primary vaccination of combined hepatitis A and B vaccine, to assess antibody persistence and a retrospective safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received GSK Biologicals' combined hepatitis A and B vaccine in the primary study (HAB-082). Subjects were aged 12 to 15 years at the time of the first vaccination.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2003-09; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Immune persistence in terms of anti-HAV and anti-HBs antibodies and GMCs, 5 and 6 years after administration of first vaccine dose. An additional dose of the study vaccine will be given (between 6 to 12 months after the Year 6 time point) to subjects who

SECONDARY OUTCOMES:
To record the SAEs that was reported since the last time point.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Australia (2):
  - GSK Investigational Site, Paramatta, New South Wales
  - GSK Investigational Site, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 100386 (EXT Y5) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100386 (EXT Y5) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100386 (EXT Y5) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 100386 are summarised with study 100387 on the GSK Clinical Study Register.
- Available data/document: Clinical Study Report: 100386 (EXT Y5) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100386 (EXT Y5) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register